CLINICAL TRIAL: NCT04779697
Title: GLP-1 Analogue Effects on Food Cues, Stress, Motivation for Highly Palatable Foods, and Weight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2000027868; 2R01DK099039-06 (NIH)
Record Dates: First submitted 2021-02-10; First posted 2021-03-03 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GLP-1a (Experimental): GLP-1a Semaglutide target dose of 1.2 mg administered weekly over 12 weeks
  Interventions: Drug: GLP-1 analogue - semaglutide
- Placebo (Placebo Comparator): Placebo pen administered weekly over 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GLP-1 analogue - semaglutide — GLP-1 analogue - semaglutide - administered once weekly for a total of 12 weeks
  Other Names: Semaglutide
  Arms: GLP-1a
Other: Placebo — Placebo - administered once weekly for a total of 12 weeks
  Arms: Placebo

SUMMARY:
To examine response to a glucagon-like peptide-1 analogue vs. placebo in patients with obesity and assess impact on craving, hunger, stress, and weight outcomes.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled 12-week study with GLP-1 analogue (semaglutide) in men and women with obesity (BMI 30-49.9 kg/m2) in a validated laboratory model to identifying processes underlying greater food craving, intake and weight change, in order to test mechanisms by which a GLP-1 analogues may exerts significant weight effects in obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI ranging from 30-49.9 kg/m2
* No significant medical problems, including diabetes
* No history of HgbA1c <6.5%
* English speaking and able to read English and complete study evaluations
* Able to provide informed written and verbal consent

Exclusion Criteria:

* Any significant current medical conditions, including neurological, renal, thyroid, cardiovascular, liver, endocrine or immune conditions, including diagnosis of T2DM or T1DM by American Diabetes Association (ADA) criteria
* Meet current or past DSM-IVR criteria for alcohol dependence or any substance use disorders, including nicotine, or psychiatric disorders, including eating disorders, or use of any psychiatric medications, including anxiolytics, antidepressants, naltrexone or antabuse, anti-smoking medications
* Current active participation in a weight loss program or weight loss of >10% of total body weight during the prior 6 months
* Taking any other anti-obesity medication
* History of pancreatitis, medullary thyroid cancer, or MEN syndrome, or (6) women who are pregnant or lactating, or peri/postmenopausal

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ania Jastreboff, MD, PhD, Principal Investigator — Internal Medicine (Endocrinology) and Pediatrics (Pediatric Endocrinology);; Rajita Sinha, PhD, Principal Investigator — Psychiatry; Director Yale Stress Center
Locations (1):
- The Yale Stress Center: Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GLP-1a | Placebo
Started | 48 | 48
Completed | 43 | 43
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics presented are for those that completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | GLP-1a | Placebo | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (9.4) | 36 (8.7) | 36.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 31 | 33 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 26 | 29 | 55
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 86
Years of Education [Mean (Standard Deviation); unit: years] | 16.1 (2.3) | 16.4 (2.7) | 16.3 (2.5)
Regularly Use Substances [Count of Participants; unit: Participants]
  Yes | 21 | 13 | 34
  No | 22 | 30 | 52
Baseline Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 37.3 (4.5) | 36.9 (4.2) | 37.1 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Craving Score
Description: Change in craving score will be measured using a validated and revised questionnaire called Food Craving Inventory (FCI-R). FCI-R is an 28-item questionnaire that measures how often participants experienced specific food cravings for each of 28 different food types. Participants can respond to each item from "not at all" (score=1) to "more than ever" (score=5), with total FCI-R score range of 28-140. Higher mean scores indicate greater average food craving. A negative change indicates a decrease in craving with treatment.
Time Frame: Average change in avg FCI craving score from week 0 to end of treatment (week 12) computed as avg FCI score at week 12 - avg FCI score at Week 0.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | GLP-1a | Placebo
Number analyzed (Participants) | 43 | 43
score | -0.7 (0.6) | -0.3 (0.4)
Statistical Analysis 1: Comparison: GLP-1a vs Placebo; Test type: Superiority; p < 0.001, ANOVA

2. Primary Outcome: Change in Hunger Score
Description: Hunger will be measured in a Visual Analog Scale (VAS) range from 0 to 10. Higher VAS indicates greater hunger. Negative change in score indicates less hunger with treatment.
Time Frame: Average change in hunger VAS rating from week 0 and end of study week 12 (week 12 VAS - Week 0 VAS)
Population: Data presented here is for all participants that completed the assessment.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | GLP-1a | Placebo
Number analyzed (Participants) | 40 | 38
score | -0.5 (1.7) | -0.1 (1.7)
Statistical Analysis 1: Comparison: GLP-1a vs Placebo; Test type: Superiority; p > 0.27, ANOVA

3. Primary Outcome: Change in Food Intake
Description: Food intake will be measured in total calorie energy density during a validated observed laboratory task called the Food Snack Test (FST).Negative change indicates a lower food intake with treatment.
Time Frame: Change in FST total calorie energy density (totalcalED)from FST at week 0 and FST during treatment at week 12 (week 12 FST - Week 0 FST totalcalED change)
Population: Data presented here is for all participants that completed the assessment.
Measure: Mean (Standard Deviation); unit: Kcalories
Arm/Group | GLP-1a | Placebo
Number analyzed (Participants) | 40 | 38
Kcalories | -0.4 (1.8) | 0.4 (2.4)
Statistical Analysis 1: Comparison: GLP-1a vs Placebo; Test type: Superiority; p < 0.043, ANOVA; Model includes a gender interaction term

4. Secondary Outcome: Change in Food Intake - Real-World
Description: Food intake will be measured in Kcalories using 3-day 24hr recall (ASA24). A negative change indicates lower food intake with treatment.
Time Frame: Average change from baseline to end of treatment (Kcalories at week 12 - week 0)
Population: Data presented here is from all participants that completed the assessment.
Measure: Mean (Standard Deviation); unit: Kcalories
Arm/Group | GLP-1a | Placebo
Number analyzed (Participants) | 38 | 37
Kcalories | -485.7 (657.6) | -124.5 (583.5)
Statistical Analysis 1: Comparison: GLP-1a vs Placebo; Test type: Superiority; p < 0.015, ANOVA

5. Secondary Outcome: Change in Stress Score
Description: Stress, measured as total summed score on the 14-item Perceived Stress Scale, with higher scores indicating greater subjective stress. A negative change indicates lower stress with treatment. The Perceived Stress Scale (PSS)-14 has a total score range of 0 to 56, with individual items scored from 0 ("Never") to 4 ("Very often") and positively worded items reverse-scored before summing.
Time Frame: Average change in stress score from week 0 to end of treatment week 12 (Week 12 - Week 0)
Population: Data presented here is from all participants that completed the assessment.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | GLP-1a | Placebo
Number analyzed (Participants) | 36 | 40
score | -2.8 (7.2) | -1.7 (8.1)
Statistical Analysis 1: Comparison: GLP-1a vs Placebo; Test type: Superiority; p > 0.53, ANOVA

6. Other Pre Specified Outcome: Change in Weight
Description: Percent change in Weight in kilograms will be assessed using a bioimpedance scale. higher negative score indicates greater change with treatment.
Time Frame: Average Weight Change from baseline week 0 to end of treatment week 12 (Week 12 - week 0)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GLP-1a | Placebo
Number analyzed (Participants) | 43 | 43
percent change | -4.53 (4.59) | -0.17 (4.01)
Statistical Analysis 1: Comparison: GLP-1a vs Placebo; Test type: Superiority; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | GLP-1a | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/48
Other Adverse Events (participants affected / at risk) | 39/48 | 32/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLP-1a (N=48) | Placebo (N=48)
Chest Pain (General disorders) | 1 (1) | 0 (0) — Chest Pain Requiring Overnight Evaluation in ED Cardiac Observation Unit- Deemed "Muscle Strain"
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLP-1a (N=48) | Placebo (N=48)
Abdominal Pain (Gastrointestinal disorders) | 15 (31) | 10 (10)
Bloating/Gas (Gastrointestinal disorders) | 5 (12) | 3 (4)
Constipation/Hard Stools (Gastrointestinal disorders) | 9 (11) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 14 (26) | 5 (10)
Gastroesophogeal Reflux (Gastrointestinal disorders) | 9 (17) | 1 (3)
Lack/Loss of Appetite (Gastrointestinal disorders) | 6 (8) | 3 (3)
Nausea (Gastrointestinal disorders) | 28 (75) | 10 (15)
Vomiting (Gastrointestinal disorders) | 13 (28) | 2 (2)
Chills (General disorders) | 5 (5) | 1 (1)
Fatigue (General disorders) | 7 (9) | 3 (3)
Fever (General disorders) | 5 (5) | 0 (0)
Injection Site Reaction (General disorders) | 5 (5) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 4 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 4 (9) | 1 (1)
Headache/Migraine (Nervous system disorders) | 14 (26) | 9 (16)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Sore Throat/Throat Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT04779697/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04779697/ICF_001.pdf